CLINICAL TRIAL: NCT04486183
Title: Effects of Different Methods Used to Take Blood Samples on Blood Glucose Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Eda Ergin, Asistant Professor,Department of Fundamentals Nursing,, Izmir Bakircay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Eda ERGIN, PhD,RN; Ayten Zaybak (Other: Ege University, Turkey, İzmir)
Record Dates: First submitted 2020-07-14; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Blood Glucose, Low
Keywords: Blood Glucose Measurements; Venous Blood; Capillary Blood

STUDY DESIGN:
Intervention Model Description: This was a quasi-experimental study with a single group and simultaneous (matched) sample conducted with the purpose of examining whether or not there is a difference between venous and capillary blood samples in blood glucose level measurements and the effects of different methods used in skin cleaning before collecting blood samples on measurement results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The data were collected by the researcher at the waiting room of the blood collection unit at a close distance to the lavatory. The capillary first and second blood drop values taken from the patients after fasting and at two hours following OGTT and capillary and venous blood glucose values were compared.
  Interventions: Other: capillary blood samples

INTERVENTIONS:
Other: capillary blood samples — The patient's finger was wiped with alcohol, left to dry, and the first and second blood drops were read The patient was asked to wash their hands, their finger was perforated with a strip, and the first and second blood drops were read The finger of the patient whose hands had been washed was wiped with alcohol, left to dry, and the first and second blood drops were read Venous blood was collected for blood sugar measurement 2 hours after the patient had a beverage containing 75 gr sugar for OGTT The patient was ensured to wash their hands, their finger was wiped with alcohol, and the first and second blood drop glucose values were measured and recorded
  Other Names: capillary blood samples were taken from the same participant in four different ways

SUMMARY:
Aims and Objectives: The purpose of this study is to compare whether or not there is a difference between venous and capillary blood samples in blood glucose measurements and investigate the effects of different aseptic methods used in skin cleaning before collecting blood samples on measurement results.

Background: Capillary blood glucose measurement is a frequently used measurement method in both clinical environments and the home environment. However, several different aseptic techniques are used in collecting blood samples for glucose measurement.

Design and Methods: This was a quasi-experimental study that was conducted with 109 patients who visited the blood collection unit of a University Hospital located in Western Turkey for 75 gr OGTT between November 2017 and April 2018. The capillary first and second blood drop values taken from the patients after fasting and at two hours following OGTT and capillary and venous blood glucose values were compared.

DETAILED DESCRIPTION:
The data were collected by the researcher at the waiting room of the blood collection unit at a close distance to the lavatory. A nurse working at the venous blood sample unit collected fasting and 2 hours after OGTT venous blood samples from the individuals who arrived at the blood collection unit for 75 gr OGTT. All venous blood and capillary blood samples were obtained in a shorter time than 5 minutes. In this study, capillary blood samples were taken from the same participant in four different ways:

* As the first intervention, the middle finger of the individuals agreeing to participate in the study was rubbed and wiped with a cotton infused with 70% alcohol, and 10 seconds were given for it to dry. Afterwards, by perforating the finger with a lancet, firstly the first blood drop glucose value and then the second blood drop glucose value were measured.
* As the second intervention, after ensuring that the individuals washed their hands with soap at the lavatory of the blood collection unit and dried their hands with paper towels, the middle finger of the right hand was rubbed, perforated with a lancet, and firstly the first blood drop glucose value and then the second blood drop glucose value were measured.
* As the third intervention, for the individuals whose hands had been washed, the middle finger of the left hand was rubbed and wiped with 70% alcohol-infused cotton, and 10 seconds were given for it to dry. The finger was perforated with a lancet and the first and second blood drop glucose values were recorded.
* As the fourth intervention, 2 hours after the individuals drank a beverage containing 75 gr of sugar for OGTT, in a state where their hands had been washed, the finger was wiped with 70% alcohol, left to dry, perforated with a lancet, and the first and second blood drop glucose values were measured and recorded

ELIGIBILITY:
Inclusion Criteria:

* who had both upper extremities,
* good capillary saturation,
* blood glucose monitoring requests for OGTT,
* who were fasting for 8-12 hours before giving blood,
* who had requests for 75 gr sugar loading
* who volunteered to participate in the study.

Exclusion Criteria:

* who refused to participate in the study,
* whose capillary blood glucose could not be looked at after sugar loading.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | at 6-month
  10 questions on the sociodemographic characteristics of the participants such as age, sex, height-weight, status of DM diagnosis in the family, status of having another chronic disease and status of smoking and alcohol consumption
Data Record Form | at 6-month
  The individuals' venous blood glucose values, capillary fasting blood glucose first and second blood drop values measured with aseptic techniques and the first and second blood drop values of the venous and capillary blood glucose 2 hours after OGTT were recorded into a "Data Record Form". As the glucometer device in the study, Roche's Accu-Chek® Performa Nano brand measurement device was used

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Bakırçay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ergin E, Zaybak A. Effects of Different Methods Used to Take Blood Samples on Blood Glucose Measurements. Clin Nurs Res. 2022 Jan;31(1):29-38. doi: 10.1177/10547738211024782. Epub 2021 Jul 5. PMID 34218680